CLINICAL TRIAL: NCT06682455
Title: Deciphering AMD by Deep Phenotyping and Machine Learning- Prospective Study - SUMMIT (Part 2)
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Southampton (Other)
Collaborators: King's College London (Other); Imperial College London (Other); Medical University of Vienna (Other); University of Michigan (Other); University College, London (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 256931; 47270 (Other: University of Southampton)
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with diagnosed intermediate age-related macular degeneration

SUMMARY:
We will conduct a prospective, non-interventional roll-over extension of the PINNACLE study (Deciphering AMD by deep phenotyping and machine learning). This will include up to 300 intermediate AMD participants (= approximately 450 untreated intermediate AMD eyes, including both unilateral (AREDS IV) and bilateral (≥AREDS II)). As per the PINNACLE study, SUMMIT study participants will continue to be followed using OCT imaging every 4 months for a further 2-years, to specifically investigate the morphological sequence of events preceding the conversion towards late AMD. Across both studies combined, we will be able to detect the earliest focal sites of disease progression over a total 5-year follow-up.

DETAILED DESCRIPTION:
Participants who have taken part in the PINNACLE study and have progressed to the final visit (i.e. have not made the decision to withdraw or met any withdrawal criteria prior to completing month 36/visit 10), within 12 months of enrolment to SUMMIT will be considered for this cohort.

We will recruit patients with a continued diagnosis of 1) intermediate AMD in the study eye and advanced AMD in the non-study eye or 2) patients with bilateral intermediate AMD (where both eyes will be included).

As within PINNACLE, there will be four clinical sites performing detailed assessments on their recruited patients, and an additional eight referral sites in the United Kingdom who will follow patients by Spectral Domain Optical Coherence Tomography (SD-OCT) every 4 months. The acquired images from all sites will be sent to the Vienna Reading Centre for review.

After consent, study assessments including both structural and functional visual testing and imaging procedures, and the collection of medical and medication data will be performed at 4-monthly intervals across a maximum 2-year period. Participants will attend a maximum of 6 visits, 2 of which (M48 and M60), will be classified as 'annual' visits, where enhanced imaging and testing will take place to further identify and assess focal and global changes.

Demographic data collected as part of the PINNACLE study baseline procedures, including birth year, smoking history and body mass index data will not be re-collected as part of the SUMMIT study. The information previously collected will however be included within the SUMMIT analysis, as has also been considered previously. The data extracted from the genotyping samples within the PINNACLE study will also be included in the SUMMIT final analysis, but no additional samples or research on existing samples will be performed under the SUMMIT study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Have taken part in the PINNACLE study and progressed to/completed the final M36/V10 study visit.
2. Have not been considered 'withdrawn' (either by 'opt-out', or any reason that would deem them ineligible, e.g. disease progression) from the PINNACLE study at any timepoint.
3. Have a period of no longer than 12 months between their final M36/V10 PINNACLE study visit and the first SUMMIT study visit (if M36/V10 was missed, the participant will still be eligible if M32/V9 completion date is within 12 months of enrolment).
4. Continued diagnosis of intermediate AMD (as defined by Ferris et al PMID: 23332590) in both eyes (i.e. large drusen > 125 µm and/or any definite hyper- or hypopigmentary abnormalities associated with medium or large drusen), or intermediate AMD as defined above in one eye (study eye) and advanced AMD (GA or MNV secondary to AMD) in the other eye.

   Participants enrolled with both eyes (OU) on the PINNACLE study, will still be eligible to enrol under OD/OS only, should one eye have been withdrawn prior to completing PINNACLE, or considered no longer eligible during enrolment on SUMMIT.
5. Have media clarity and pupillary dilation for adequate imaging and functional tests.
6. Deemed able to meet the physical demands of attending 4-monthly appointments and undergo the examinations as listed in section 7.3, for the study duration (maximum 2 years).

Exclusion Criteria:

1. Co-existent ocular disease, which might affect visual function or retinal morphology.
2. Established glaucoma in either study eye or fellow eye with evidence of visual field loss or retinal nerve fibre loss (ocular hypertension is not an exclusion criterion unless associated with visual field loss or retinal nerve fibre loss in either eye).
3. Cataract sufficient to affect retinal imaging.
4. Myopia > minus 6 diopters or a history of myopia > minus 6 diopters if patient has had cataract/refractive surgery.
5. Major ocular surgery (e.g. corneal transplant, vitreo-retinal surgery) 3 months prior or anticipated within the next 6 months following enrolment (not including cataract surgery).
6. Taking drugs known to cause retinal toxicity, such as hydroxychloroquine or tamoxifen.
7. OCT evidence of MNV (e.g sub-retinal scar tissue, sub-retinal fluid or intra-retinal fluid associated with a pigment epithelial detachment).
8. Participants who have completed the PINNACLE study >12 months prior to their enrolment on SUMMIT.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have completed the PINNACLE study (Part 1) and have; 1) intermediate AMD in the study eye and advanced AMD in the non-study eye or 2) patients with bilateral intermediate AMD (where both eyes will be included).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity / specificity of OCT biomarkers | 2 years
  Sensitivity / specificity of OCT biomarkers identified in the retrospective branch of our study at predicting disease progression towards advanced AMD i.e. development of early onset neurosensory atrophy or choroidal neovascularisation.

SECONDARY OUTCOMES:
Sensitivity / specificity of novel imaging characteristics | 2 years
  Sensitivity / specificity of novel imaging characteristics e.g. fundus autofluorescence, AO-OCT, OCT-A at predicting disease progression; ROC curves; time from development of imaging change to development of these end-points; structure-function correlation; structure-genotype correlation; predictive risk models.

CONTACTS AND LOCATIONS:
Locations (8):
- Medical University of Vienna, Vienna, Austria
- United Kingdom (7):
  - The Princess Alexandra Hospital Nhs Foundation Trust, Harlow, Essex
  - University Hospital Southampton, Southampton, Hampshire
  - St Mary's Hospital, Newport, Isle Of Wight
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - Frimley Health Nhs Foundation Trust, Frimley, Surrey
  - Salisbury Nhs Foundation Trust, Salisbury, Wiltshire
  - Moorfields Eye Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Requests to access anonymised Individual Participant Data (IPD) can be made on application to the Trial Management Group Data Access Committee.
Supporting Information: Study Protocol, SAP
Time Frame: Currently available and can be accessed indefinitely.
Access Criteria: Requests for further information such as a clinical study report will be considered by the investigators following the end of the study and publication of primary outputs.